CLINICAL TRIAL: NCT05649449
Title: Money Follows the Person Through Self-Directed Care in Florida
Brief Title: Testing Self-Directed Care in Florida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith A. Cook, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY2008-0970
Record Dates: First submitted 2022-12-05; First posted 2022-12-14 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Mental Disorder
Keywords: self-directed care
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Self-directed care is a recovery-oriented model of community mental health service delivery in which participants manage a personal budget from which they purchase goods and services, including specific types of mental health care, social supports, and items that allow them to recover their health and emotional wellness and live independently.
Who Masked: Outcomes Assessor
Masking Description: Research interviewers are blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants meet with self-directed care program staff called brokers to receive a program orientation, share perceptions of their current life situation and mental health status, and review past year behavioral health service use as well as participants' views of service helpfulness. This culminates in participants' choice of recovery goals and development of an individual budget to pay for for services and material goods directly related to recovery goals. After budget approval by the program supervisor, brokers make purchases. At quarterly meetings, brokers and participants discuss the latter's progress toward recovery goals and create the next quarter's budget. After receiving 12 months of SDC services, participants are helped to transition back to usual community mental health services.
  Interventions: Behavioral: Self-Directed Care
- Control (Active Comparator): Subjects receive routine mental health care from community agencies consisting of outpatient services coordinated at community behavioral health programs.
  Interventions: Behavioral: Services as usual

INTERVENTIONS:
Behavioral: Self-Directed Care — Participants meet with self-directed care program staff called brokers to receive a program orientation, share perceptions of their current life situation and mental health status, and review past year behavioral health service use as well as participants' views of service helpfulness. This culminates in participants' choice of recovery goals and development of an individual budget to pay for for services and material goods directly related to recovery goals. After budget approval by the program supervisor, brokers make purchases. At quarterly meetings, brokers and participants discuss the latter's progress toward recovery goals and create the next quarter's budget. After receiving 12 months of SDC services, participants are helped to transition back to usual community mental health services.
  Arms: Experimental
Behavioral: Services as usual — Participants receive usual outpatient psychiatric care delivered at community programs from which the person can choose from an array of services negotiated with the state mental health authority.
  Arms: Control

SUMMARY:
This study tests a psychosocial intervention called mental health self-directed care by assessing its impact on recovery, mental health status, rehabilitation outcomes, and service costs in the state of Florida.

DETAILED DESCRIPTION:
With additional funding from the National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR), a new cohort of 40 study subjects will be recruited in the state of Florida to test mental health self-directed care (SDC). SDC is a self-directed model of service delivery in which participants manage a personal budget from which they purchase goods and services, including specific types of mental health care, social supports, and items that allow them to recover their health and emotional wellness and live independently. Investigators are studying the impact of SDC on recovery, mental health status, rehabilitation outcomes, and service costs. Working with Lutheran Services Florida, a public managing entity coordinating mental health care management in northeastern and central Florida, adults with mental health conditions will be recruited into the study and randomly assigned to receive SDC for one year or continue receiving services as usual. Assessments will occur at baseline, 6- and 12-month followup.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Serious mental illness
* Receiving services coordinated by behavioral health managing entity

Exclusion Criteria:

* Cognitive impairment preventing informed consent
* Enrollment in Medicaid/Medicare
* Representative payeeship
* Court-mandated treatment
* Recent substance disorder crisis
* In residential treatment
* History of violent behavior in the past 10 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Change in perceived competence for mental health self-management | study entry (pre-intervention), 6-months (intervention mid-point), 12-months (immediate post-intervention)
  Perceived competence is measured with the Perceived Competence Scale that includes 4 items that assess subjects' self-rated ability to manage their mental health and recovery, with scores ranging from 4 to 28, with higher scores indicating greater perceived competence for mental health self-management.

SECONDARY OUTCOMES:
Change in met and unmet needs related to multiple life domains | study entry (pre-intervention), 6-months (intervention mid-point), 12 months (immediate post-intervention)
  Change in met and unmet needs is measured with the Camberwell Assessment of Need Short Appraisal Schedule with 22 items that assess needs across multiple life domains such as psychological distress, general health, and finances, which results in 2 scores, each ranging from 0-22, with higher scores indicating more met needs or more unmet needs.
Change in perception of service providers as supportive of client autonomy | study entry (pre-intervention), 6-months (intervention mid-point), 12-months (immediate post-intervention)
  Change in provider support for client autonomy is measured by the Health Care Climate Questionnaire with 6 items that assess the degree to which subjects rate their services providers as encouraging autonomy by providing information, encouraging choice, and acknowledging subjects' emotions, with scores ranging from 6 to 42, with higher scores indicating more perceived autonomy support.
Change in self-rated recovery from mental illness | study entry (pre-intervention), 6-months (intervention mid-point), 12-months (immediate post-intervention)
  Change in self-rated recovery is measured by the Recovery Assessment Scale with 41 items that assess perceived level of recovery from mental illness, with higher scores indicating greater recovery.
Change in employment status | study entry (pre-intervention), 6-months (intervention mid-point), 12-months (immediate post-intervention)
  Assessment of employment status using the U.S. Bureau of Labor Statistics definition of paid employment which ranges from 0 (no) to 1 (employed) where a higher score indicates employment.
Change in service costs | 12-month period of study participation
  Service cost is measured by the dollar amount of reimbursement paid by the behavioral health managing entity to a service provider or program for a paid claim for a discrete service with scores ranging from 0 dollars to no upper limit of dollars where higher scores indicate greater cost.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Department of Psychiatry, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No